CLINICAL TRIAL: NCT02686801
Title: Determinants of Body Composition at Discharge and Fat-Free Mass as an Indicator of Neurological Development at 2 Years in Very Preterm Infants : OPTIPREMA Study
Brief Title: Body Composition at Discharge and Neurological Development at 2 Years in Very Preterm Infants (OPTIPREMA)
Acronym: OPTIPREMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital de la Croix-Rousse (Other)
Responsible Party: Principal Investigator, Jean-charles PICAUD, MD, PhD, Professor of pediatrics, Hôpital de la Croix-Rousse
Other Study IDs: OPTIPREMA
Record Dates: First submitted 2016-02-02; First posted 2016-02-22 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Premature Birth of Newborn
Keywords: nutrition; prematurity; body composition
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the perinatal factors influencing body composition at discharge in very preterm infants and the relationship between fat free mass and further neurocognitive development.

DETAILED DESCRIPTION:
Postnatal growth is a crucial in premature infants as it could be correlated with the long-term cognitive development. Recent data from the literature show that it is possible - with appropriate nutritional care - to reduce the initial weight loss and to ensure that the growth deficit accumulated is then less important than was previously observed. The quantitative objective is to achieve growth that is at least equivalent to that of the fetus (12-18 g/kg.day according to postconceptional age). Children often grow slowly during the first 10 days of life, so they accumulate a growth deficit that should be compensated secondarily. Therefore, optimum postnatal growth is 20 g/kg.day, rather than 15 g/kg.day. It is also important to assess the quality of growth, particularly fat free mass. The objective of nutritional care is dual: a sufficient weight gain (close to fetal growth rate) but also a relevant body composition. However, there is very little data on body composition of premature babies at discharge. It is now possible to measure quickly (one minute), simply and noninvasively using pediatric air-displacement plethysmography. Previous studies using more complex search techniques to implement (dual energy X-ray absorptiometry) showed excessive body fat at discharge in premature babies. Reference values collected using pediatric air-displacement plethysmography were published in 2011. Nutritional practices and strategies have significantly evolved in the past years to support such objectives: improvement of early parenteral nutrient intake, new fortifiers for human milk, new preterm formulas and early beginning of enteral nutrition. Individualized fortification of human milk helps to provide preterm infants with sufficient amount of nutrients. The modern nutritionnal care in preterm infants results in earlier and higher protein and energy intakes than previously performed. It improves some anthropometric parameters but little is know about body composition at discharge. Furthermore, exposition to high nutrients intake could lead to metabolic and hormonal imprinting with an increased risk of diabetes and cardio-vascular diseases in adulthood.

OPTIPREMA aim to focus the link between nutrient intakes during hospitalization, body composition at discharge and relationship between fat free mass variations at discharge and neurodevelopment at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns (less or equal to 32 weeks gestation and / or birthweight less or equal to1500g).
* Admitted in the Neonatal unit before day-of-life 7, staying at least 15 days in the unit, and discharged home at ≥ 35 weeks postconceptional age directly from the neonatal unit (no transfer)
* Oral Parental consent

Exclusion Criteria:

* Hemodynamic or cardiovascular instability requiring continuous monitoring or perfusion, incompatible with pediatric air-displacement plethysmography
* Pathology inducing neurodevelopment troubles
* Transfer in an other hospital before discharge
* Hemodynamic or cardiovascular instability requiring continuous monitoring or perfusion, incompatible with pediatric air-displacement plethysmography

Ages: 1 Week to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Fat free mass at discharge | pediatric air-displacement plethysmography measurement will be done at 36 to 40 weeks postconceptional age
  Fat-fee mass percentage at discharge by pediatric air-displacement plethysmography After checking inclusion and non-inclusion criteria and obtaining oral informed consent from newborn legal authority or parents, pediatric air-displacement plethysmography is performed in the last week of hospitalization. Body composition estimation is completed by clinical and demographic data collection and collection of information about neonatal nutrition.

SECONDARY OUTCOMES:
Factors (clinical characteristics at birth and morbidity, feeding regimen) influencing body composition at discharge | pediatric air-displacement plethysmography will be done at 36 to 40 weeks postconceptional age
  Factors (nutritional and others) influencing body composition of preterm infants (<35 weeks gestation) at discharge. Analysis will focuss on condotions that could be influenced by neonatal care, such as weight gain.
Prediction of fat free mass at discharge | pediatric air-displacement plethysmography will be done at 36 to 40 weeks postconceptional age
  Prediction of fat free mass at discharge from anthropometric data, nutritional intakes, and evolution during hospitalization.
Anthropometric parameters at discharge and at 2 years | measurements will be done at 36 to 40 weeks postconceptional age and at 2 years of age
  Relationship between anthropometric parameters and body composition at discharge and growth at 2 years
Body mass index at discharge and at 2 years | measurements will be done at 36 to 40 weeks postconceptional age and at 2 years of age
  Relationship betwen body mass index as an marker of body composition at discharge and growth at 2 years
Fat free mass in preterm infants fed human milk fortified in an individualized way | pediatric air-displacement plethysmography will be done at 36 to 40 weeks postconceptional age
  Impact of optimized feeding regimen using adjustable individualized fortification of human milk on fat free mass at discharge
Developmental score as measured by an appropriate neurodevelopmental test at 2 years | Neurodevelopmental assessment at 2 years old
  Children neurological development at 2 years old evaluated according to the follow-up routine evaluation or very low birth weight infants

CONTACTS AND LOCATIONS:
Overall Officials: jean-charles picaud, MD, PhD, Principal Investigator — Hopital de la croix rousse
Locations (1):
- Hopital de la croix rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Larcade J, Pradat P, Buffin R, Leick-Courtois C, Jourdes E, Picaud JC. Estimation of Fat-free Mass at Discharge in Preterm Infants Fed With Optimized Feeding Regimen. J Pediatr Gastroenterol Nutr. 2017 Jan;64(1):115-118. doi: 10.1097/MPG.0000000000001261. PMID 27149252